CLINICAL TRIAL: NCT00003565
Title: A Study of Population Pharmacokinetics of Docetaxel (Taxotere) in Caucasian and African-American Cancer Patients
Brief Title: Docetaxel in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9871; U10CA031946 (NIH); CALGB-9871; CDR0000066631 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Cancer; Breast Cancer; Head and Neck Cancer; Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage IV nasopharyngeal cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; pulmonary carcinoid tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel (Experimental): OUTLINE: Patients receive docetaxel IV over 1 hour on day 1. Patients may receive additional courses beginning 21 days after the first docetaxel dose at the discretion of the physician.
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to compare the effectiveness of docetaxel in treating Caucasian and African American patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the population pharmacokinetics of docetaxel in Caucasians and African American patients with solid tumors.
* Compare the pharmacodynamic effect of a single dose of docetaxel in relation to hematological toxicity in these patient populations.
* Determine the CYP3A4 genotype and P-glycoprotein (P-gp) expression and their relationship to docetaxel clearance in these patient populations.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1. Patients may receive additional courses beginning 21 days after the first docetaxel dose at the discretion of the physician.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unresectable solid tumors (e.g., lung, breast, head and neck, bladder)
* Clinically suitable for treatment with single agent docetaxel
* Caucasian (at least 2 generations originating in any of the original peoples of Europe, North Africa, or the Middle East) OR
* African American (at least 2 generations originating in any of the black racial groups of Africa)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 1.5 times ULN AND
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* BUN no greater than 1.5 times ULN
* Creatinine no greater 1.5 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation

Chemotherapy:

* No prior docetaxel
* Prior paclitaxel allowed
* 1 or 2 prior chemotherapy regimens allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormones for disease related conditions
* Concurrent steroids for adrenal failure allowed

Radiotherapy:

* At least 2 weeks since prior radiotherapy
* Palliative radiotherapy allowed except whole brain irradiation for CNS disease

Surgery:

* Not specified

Other:

* At least 48 hours since prior or concurrent ethanol (CYP3A enzyme inducer) or grapefruit juice (CYP3A enzyme inhibitor)
* At least 7 days since prior or concurrent CYP450 inducing drugs:

  * Antiseizure medications: phenobarbital, phenytoin, carbamazepine, or lamotrigine
  * Anti-TB therapy: rifampin, isoniazid, or sulfinpyrazone
* At least 7 days since prior or concurrent CYP450 3A inhibiting drugs:

  * Macrolides: erythromycin, clarithromycin, azithromycin, or roxithromycin
  * Azoles: ketoconazole, fluconazole, or itraconazole
  * Other antibiotics: metronidazole or chloramphenicol
  * Anti-HIV drugs: ritonavir, indinavir, nelfinavir, or delavirdine
  * Immunosuppressive agents: cyclosporine
  * Antidepressant agent: nefazodone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 1998-09; Primary Completion 2006-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Lewis, MD, Study Chair — Norris Cotton Cancer Center
Locations (74):
- United States (72):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- McGill University, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Lewis LD, Miller AA, Rosner GL, Dowell JE, Valdivieso M, Relling MV, Egorin MJ, Bies RR, Hollis DR, Levine EG, Otterson GA, Millard F, Ratain MJ; Cancer and Leukemia Group B. A comparison of the pharmacokinetics and pharmacodynamics of docetaxel between African-American and Caucasian cancer patients: CALGB 9871. Clin Cancer Res. 2007 Jun 1;13(11):3302-11. doi: 10.1158/1078-0432.CCR-06-2345. PMID 17545536